CLINICAL TRIAL: NCT00549237
Title: Perioperative Nutrition in Gastric Bypass Surgery for Morbid Obesity
Brief Title: Perioperative Nutrition in Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER 07 - 096
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Complications; Gastric Bypass
Keywords: RYGBP; Early nutrition; Lean body mass; Length of stay; Body Composition
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition (Active Comparator): Pre-operative Glucose load and post-operative immediate enteral nutrition
  Interventions: Dietary Supplement: Glucose load (Nutricia); Other: Post operative early enteral feeding
- Control (No Intervention): No pre-operative glucose load. No early post-operative nutrition

INTERVENTIONS:
Dietary Supplement: Glucose load (Nutricia) — Pre-operative glucose load: 800 ml of PreOp (Nutricia) 12 h before surgery; 400 ml of PreOp (Nutricia) 2 hours before surgery
  Other Names: PreOp, Nutricia
  Arms: Nutrition
Other: Post operative early enteral feeding — Enteral feeding starting 6 hours post surgery
  Arms: Nutrition

SUMMARY:
The aim of this study is to demonstrate the influence of peri-operative nutrition on the preservation of lean body mass after gastric bypass, as well as it's influence on postoperative complications.

DETAILED DESCRIPTION:
Outcome measures:

* Lean body mass
* Length of hospital stay
* Weight loss
* Postoperative complications
* Cost

ELIGIBILITY:
Inclusion Criteria:

* RYGBP surgery planned
* Age over 18
* Informed consent

Exclusion Criteria:

* Previous bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Post-operative body mass composition | 2 years

SECONDARY OUTCOMES:
Post-operative complications | 30 days
Length of stay | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan E Azagury, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires Genève, Geneva, Canton of Geneva, Switzerland